CLINICAL TRIAL: NCT01152801
Title: A Phase Ib, Multi-center, Open-label Study to Evaluate the Safety of RAD001 in Chinese Patients With Metastatic Renal Cell Cancer Who Are Intolerant of or Who Have Progressed Despite Treatment With VEGF-targeted Therapies
Brief Title: Safety of RAD001 in Chinese Patients With Metastatic Renal Cell Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001L2101; Chinese HA - 2008L09346 (Registry Identifier: Chinese HA)
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2014-06

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: mRCC,; everolimus,; mTOR,; intolerant of VEGF-therapies
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Everolimus

ARMS (1):
- RAD001 (Experimental)
  Interventions: Drug: Everolimus (RAD001)

INTERVENTIONS:
Drug: Everolimus (RAD001)

SUMMARY:
This is an open-label, multi-center study to evaluate the safety of RAD001 in Chinese patients with metastatic renal cell cancer who are intolerant of or have progressed despite treatment with vascular endothelial growth factor (VEGF)-targeted therapies. All patients will be treated with RAD001 10 mg daily until tumor progression (determined according to the Response Evaluation Criteria In Solid Tumors (RECIST) Criteria), unacceptable toxicity, death or discontinuation from the study for any other reason. At least 60 patients will be enrolled in the study. Screening and baseline evaluations will be performed within 28 days of the date when the patient signs the informed consent form. Baseline evaluations will be performed within two weeks of the first dose of RAD001. Screening and baseline evaluations will be performed to determine if patient meets all inclusion and exclusion criteria. All eligible patients should be enrolled in the study and will receive the first dose of RAD001 (10 mg daily) on Day 1, Cycle 1. Subsequently, patients will be asked to come to the clinic every month to complete the protocol-specified evaluations. A treatment Cycle consists of 28 days. After discontinuation of treatment with RAD001, patients will have a safety follow-up performed 28 days after the last dose of RAD001. Patients must continue with survival assessments which will be performed every 3 months from the last dose of RAD001 until up to 2 years after the last patient's first visit date.

An interim analysis focusing on safety data and a final analysis of all data are planned. All patients still receiving the study drug at the time of the final analysis will be given the option to continue treatment with RAD001 until the occurrence of unacceptable toxicity or disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Chinese origin who are ≥ 18 years old.
* Patients with histologically or cytologically confirmed metastatic renal cell carcinoma.
* Patients who are intolerant of or who have progression on or after stopping treatment with VEGF-targeted therapies within 6 months. Note: Prior treatment with vaccine therapy in the adjuvant setting and prior treatment with cytokines (i.e., IL-2, Interferon) or chemotherapy is permitted.
* Patients with at least 1 measurable lesion determined according to the RECIST Criteria Guidelines.
* Patients with history of brain metastasis who are clinically judged by the investigator as neurologically stable following definitive radiation or surgery and do not require corticosteroids may be enrolled in the study.
* Patients with a Karnofsky Performance Status ≥ 70%.
* Patients with adequate bone marrow function defined as ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hgb >9 g/dL.
* Patients with adequate liver function defined as serum bilirubin ≤ 1.5 x ULN, ALT and AST ≤ 2.5x ULN. Patients with known liver metastases who have an AST and ALT ≤ 5x ULN.
* Patients with adequate renal function which is defined as serum creatinine ≤ 2 x ULN.
* Women of childbearing potential must have had a negative serum pregnancy test within 14 days prior to the administration of RAD001.
* Patients must give written informed consent according to local guidelines

Exclusion Criteria:

* Patients who have received chemotherapy, immunotherapy, radio-therapy or any other investigational agent (including pazopanib, axitinib) within 4 weeks of study entry, or have received sunitinib® and/or sorafenib® within 2 weeks of the first dose of RAD001.
* Patients who have previously received RAD001 or other mTOR inhibitors.
* Patients with a known hypersensitivity to RAD001 or other rapamycin analogs (sirolimus, temsirolimus), or to its excipients.
* Patients who have a history of another primary malignancy ≤ 3 years, with the exception of non-melanoma skin cancer, and carcinoma in situ of uterine cervix.
* Patients receiving chronic and systemic treatment with corticosteroids or another immunosuppressive agent. Patients may receive low dose treatment of corticosteroids with a maximum dose of 20 mg prednisone or 10 mg dexamethasone per day, if they are being given for disorders such as rheumatoid arthritis, asthma, or adrenal insufficiency. Topical or inhaled corticosteroids are permitted.
* Patients with a clinically significant active bleeding diathesis.
* Patients with known HIV seropositivity, hepatitis B or C seropositivity. Patients with prior hepatitis B vaccination may be entered in the study after review of hepatitis test results by the investigator.
* Patients who have undergone major surgery within 4 weeks prior to starting study drug (e.g., intra-thoracic, intra-abdominal, or intra-pelvic), open biopsy, or significant traumatic injury, or who have not recovered from the side effects of any of the above.
* Patients with any severe and/or uncontrolled medical conditions such as: unstable angina pectoris,symptomatic congestive heart failure,myocardial infarction ≤ 6 months,serious uncontrolled cardiac arrhythmia, uncontrolled hypercholesterolemia (>300 mg/dL or 7.75 mmol/L),uncontrolled diabetes (fasting glucose > 2x ULN),an active or uncontrolled severe infection, cirrhosis, chronic or persistent active hepatitis.
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are used, they must be continued throughout the study by both sexes, and up to 8 weeks after ending treatment. Hormonal contraceptives are not acceptable as a sole method of contraception

Other protocol related inclusion/exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability profile of RAD001 (10mg daily dose) in Chinese patients who are intolerant of or have progressed on or after VEGF-targeted therapy. | 4 month + 12 month

SECONDARY OUTCOMES:
Disease control rate (DCR), best overall response rate and progression-free survival (PFS) | 12 month
Overall survival (OS) | 12 month
Systemic pre-dose exposure levels of RAD001 in Chinese patients. | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- China (5):
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai

REFERENCES:
- [Derived] Li S, Kong Y, Si L, Chi Z, Cui C, Sheng X, Guo J. Phosphorylation of mTOR and S6RP predicts the efficacy of everolimus in patients with metastatic renal cell carcinoma. BMC Cancer. 2014 May 28;14:376. doi: 10.1186/1471-2407-14-376. PMID 24886512
- [Derived] Guo J, Huang Y, Zhang X, Zhou F, Sun Y, Qin S, Ye Z, Wang H, Jappe A, Straub P, Pirotta N, Gogov S. Safety and efficacy of everolimus in Chinese patients with metastatic renal cell carcinoma resistant to vascular endothelial growth factor receptor-tyrosine kinase inhibitor therapy: an open-label phase 1b study. BMC Cancer. 2013 Mar 21;13:136. doi: 10.1186/1471-2407-13-136. PMID 23514360
- See also: Results for CRAD001L2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=12303